CLINICAL TRIAL: NCT07345091
Title: Feasibility Performance Study Protocol for ABL90 FLEX PLUS HEM
Brief Title: Feasibility Performance Study of ABL90 FLEX PLUS HEM
Acronym: ABL90FLEXHEM
Status: Recruiting | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DC-089793-ABL90FLEX-HEM-Rev3
Record Dates: First submitted 2025-09-11; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hemolysis
Keywords: IVDR; Blood Gas Analyser; In vitro diagnostic; hemolysis detection
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults, 18 years of age or older, that have been admitted to hospital and undergo blood collection: Adults, 18 years of age or older, that have been admitted to the hospital and undergo blood collection as part of their standard care will be eligible for participation. Many of these patients are admitted to the Intensive Care Unit (ICU) with acute injury or critical illness and are temporarily unconscious or sedated at the time of admission or during recovery in the intermediate care unit and post-anesthesia care unit due to their medical condition and required treatment (e.g., mechanical ventilation or sedation) and have an A- and or a V-line established for routine sample collection without additional burden as part of their standard care.
  Interventions: Diagnostic Test: The purpose of this study is to investigate the performance of the hemolysis detection function on the ABL90 FLEX PLUS HEM using arterial or venous whole blood

INTERVENTIONS:
Diagnostic Test: The purpose of this study is to investigate the performance of the hemolysis detection function on the ABL90 FLEX PLUS HEM using arterial or venous whole blood — The hemolysis detection function is a newly developed sample quality feature on the ABL90 FLEX PLUS HEM intended to detect hemolyzed samples and to improve the reliability of the results provided by blood gas analyzer.

SUMMARY:
This feasibility performance study evaluates the ABL90 FLEX PLUS HEM device for its analytical performance in a clinical setting. The study aims to evaluate the performance of the hemolysis detection feature.

DETAILED DESCRIPTION:
The study is designed to assess the feasibility and performance of the ABL90 FLEX PLUS HEM device in a clinical environment. It will involve testing whole blood samples using the device and comparing results against established reference method. The primary focus is on validating the device's performance of the hemolysis detection function. The study will be conducted at one selected clinical site with trained personnel and will follow a predefined protocol to ensure consistency and reliability of data collection. The outcomes will inform future clinical studies aimed at supporting regulatory submissions and clinical adoption.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older
* Informed consent is obtained:

  * Directly from the subject, if they are competent and able to understand the provided information and voluntarily agree to participate, or
  * If the subject is temporarily incapacitated and unable to provide informed consent at the time of sample collection, written informed consent will be obtained from the subject's legally designated representative (LDR). when the subject regains capacity after enrollment, they will be informed of study inclusion and given the opportunity to withdraw consent.
* Subject evaluated as suitable according to the protocol and for the study by the principal investigator or designee.

Exclusion Criteria:

* Subject where sample collection is evaluated by PI or designee to impose unnecessary risk.
* Subject with an invalid written informed consent or who has withdrawn consent.
* Subject with known pregnancy or who is breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, 18 years of age or older, that have been admitted to the hospital and undergo blood collection as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Percent of samples correctly classified into hemolysis bins (0-4) using ABL90 FLEX PLUS HEM hemolysis flag | At time of sample analysis (single session per sample; Day 1)
  Whole blood samples (native and contrived) are classified into five hemolysis bins based on reference ccfHb (mg/dL): bin 0 (0-100), bin 1 (101-200), bin 2 (201-400), bin 3 (401-1000), bin 4 (>1000). "Correct classification" is the proportion of samples where the ABL90 FLEX PLUS HEM hemolysis flag matches the reference bin assignment.

SECONDARY OUTCOMES:
Slope of change in ccfHb concentration over 0-45 minutes (mg/dL per minute) | 0-45 minutes after t=0 measurement (within one sample session; Day 1)
  For each sample, ccfHb is measured on ABL90 FLEX PLUS HEM at t=0, 15, 30, and 45 minutes (±5 minutes). The outcome is the slope (mg/dL/min) from linear regression of ccfHb versus time over 0-45 minutes.
Pearson correlation coefficient (r) between ABL90 ccfHb (mg/dL) and Cobas 8000 Hemolysis Index (HI) | At time of paired analysis per sample (Day 1)
  Paired measurements are obtained from the same sample: ABL90 FLEX PLUS HEM measures ccfHb (mg/dL) in S65 mode, and Roche cobas 8000 reports Hemolysis Index (HI) using the hemolysis index assay. The outcome is the Pearson correlation coefficient (r) across paired ABL90 ccfHb and Cobas HI values (unitless r).
Pearson correlation coefficient (r) between ccfHb and potassium concentration (cK+, mmol/L) after RMED aspiration manipulation | During RMED manipulation session (baseline to after 2 aspiration rounds; Day 1)
  For each sample, ABL90 FLEX PLUS HEM measures ccfHb and potassium (cK+) at baseline (no manipulation), after 1 round of RMED aspiration manipulation, and after 2 rounds. The outcome is Pearson correlation coefficient (r) between ccfHb and potassium values pooled across the three measurements (unitless r).
Percentage of native whole blood samples with hemolysis (ccfHb > 20 mg/dL) | At time of native sample analysis (Day 1)
  Among native (non-contrived) leftover arterial and venous whole blood samples, the outcome is the percentage of samples with ccfHb > 20 mg/dL as measured on ABL90 FLEX PLUS HEM.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: No